CLINICAL TRIAL: NCT03074227
Title: The FAIS-Trial: Faecal Transplantation in Adolescents With Refractory Irritable Bowel Syndrome
Brief Title: The FAIS-Trial: Faecal Microbiota Transplantation (FMT) in Adolescents With Refractory Irritable Bowel Syndrome (IBS)
Acronym: FAIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, M.A. Benninga, Prof.dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FAIS2016
Record Dates: First submitted 2017-02-28; First posted 2017-03-08 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Double-blind, randomised, placebo-controlled pilot study as well as a reversed translational part.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomised by a computerised random-number generator to one of the following two treatment arms:
  1. allogeneic faecal infusions at t=0 and t=6.
  2. autologous faecal infusions at t=0 and t=6.
  Randomisation and preparation of the faeces will be performed by one of the research assistants. He/she is the only person who will know which treatment the patient will be given and will have no role in further parts of the study.
  The randomisation list will be kept under secured access by the Clinical Research Unit of the AMC Amsterdam, who will perform the randomisation. In case of an emergency the study medication can be unblinded after consultation of the principal investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allogeneic faecal transplantation (Active Comparator): Faecal transplantation of donor stool
  Interventions: Other: Allogeneic faecal transplantation
- Autologous faecal transplantation (Placebo Comparator): Faecal transplantation of own stool
  Interventions: Other: Autologous faecal transplantation

INTERVENTIONS:
Other: Allogeneic faecal transplantation — Patients will get bowel lavage through a nasoduodenal tube. This bowel lavage consists of 2-3 litres of macrogol electrolytes (Klean-Prep) solution. After that, patients will be treated with allogeneic faecal microbiota transplantation via the nasoduodenal tube.
  Faeces will be collected from a donor.
  Other Names: FMT
  Arms: Allogeneic faecal transplantation
Other: Autologous faecal transplantation — Patients will get bowel lavage through a nasoduodenal tube at our centre. This bowel lavage consists of 2-3 litres of macrogol electrolytes (Klean-Prep) solution. After that, patients will be treated with autologous faecal microbiota transplantation via the nasoduodenal tube.Faeces will be collected from the patient him/herself, in which their own faeces (autologous) will be used as a placebo.
  Other Names: FMT
  Arms: Autologous faecal transplantation

SUMMARY:
A Double-blind randomised placebo-controlled pilot study as well as a reversed translational part To investigate whether two faecal transplantations from either allogeneic (healthy) or autologous (own) donor, administered through a nasoduodenal tube, has beneficial effects on irritable bowel syndrome (IBS) symptoms such as abdominal pain frequency and severity. Secondary objective is to study microbiota changes in faeces samples.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a chronic disorder characterized by abdominal pain or discomfort associated with a change in stool form or frequency, in the absence of a biochemical or structural explanation for these symptoms. The prevalence of IBS in the general adult population is 9.8-12.8%, which is in accordance to the prevalence of IBS in children and adolescents (6.2%-11.9%). Patients with IBS report a decreased quality of life, high work or school absence, and are more at risk than healthy controls of developing depressive and anxiety disorders. Consequently, the healthcare costs are substantial; annual costs of care for adults with IBS in the USA are estimated to be over $20 billion. Total annual costs per paediatric IBS patient in the Netherlands are estimated to be €2500. Although the pathophysiology of IBS has not been fully elucidated, pathophysiological abnormal gastrointestinal motility, visceral hypersensitivity, altered brain-gut function, low-grade inflammation, psychosocial disturbance and intestinal microbiota characteristics have been proposed to contribute to the pathophysiology. Current treatment focuses on abnormal gastrointestinal motility, altered brain-gut function and psychosocial disturbances. However, a significant amount of IBS patients has remaining symptoms, despite these treatment regimens. These patients are considered to be therapy-resistant, also called refractory. Treatment focusing on other components of the underlying pathophysiology, such as the intestinal microbiota, might therefore lead to new therapeutic successes in this group of patients. In this light, being able to modify the intestinal microbiota inrefractory IBS patients could have beneficial effects on symptoms. Faecal transplantation, a relatively new treatment regimen that enables the modification of the microbiome, has been shown to be highly effective in treating Clostridium difficile infections and also yielded promising results in patients with other diseases such as diabetes.

Objective: To investigate whether two faecal transplantations from either allogeneic (healthy) or autologous (own) donor, administered through a nasoduodenal tube, has beneficial effects on irritable bowel syndrome (IBS) symptoms such as abdominal pain frequency and severity. Secondary objective is to study microbiota changes in faeces samples.

Study design: Double-blind randomised placebo-controlled pilot study as well as a reversed translational part.

Study Population: Patients with refractory IBS, defined as a failure to improve after standard medical treatment, at least 6 sessions of a psychological therapy and absence of response to at least 1 pharmacological agent (aged 16-21 years, male/female, no concomitant medication, non-smoking), will be recruited by their (paediatric) gastroenterologist at the Academic Medical Centre (Amsterdam, the Netherlands) and patients from other hospitals will be enrolled. Donors: relatives or volunteers will serve as faeces donor, potential donors will be thoroughly screened.

Treatment: After bowel lavage with Klean-Prep, patients will be treated with faecal transplantation at t=0 and t=6 weeks, processed for duodenal tube infusion. Faeces will be collected from a healthy donor (allogeneic) as well as the patient him/herself (autologous), in which their own faeces will be used as a placebo.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Age 16-21 years
* Non-smokers
* Ability to give informed consent
* Established irritable bowel syndrome diagnosis according to the Rome IV criteria for children or adults
* According to a recently published guideline by the Rome Foundation for the design of pharmacological clinical trials in adolescents, patients are required to have an average daily pain rate of at least 30mm on the pain component scale of the IBS-SSS
* Symptoms are present for ≥12 months
* The patient has received adequate explanation and reassurance for his/her symptoms
* Appropriate dietary interventions have occurred, including the normalisation of the insoluble fibre intake and a decrease in gas producing foods
* Absence of response to a minimum of six sessions of psychological treatment (i.e. cognitive behavioural therapy and/or hypnotherapy)
* Absence of response to an adequate dose of at least one IBS specific pharmacological agent tried for a minimum of 6 weeks (like Mebeverine or peppermint oil capsules)

Donors

* Age ≥18 years
* Non-smokers
* Ability to give informed consent
* BMI 18-25 kg/m2
* Regular stool pattern

Exclusion Criteria:

Patients

* Current treatment by another health care professional for abdominal symptoms
* Known concomitant organic gastrointestinal disease
* Known diagnosis of inflammatory bowel disease (i.e. Crohns disease or ulcerative colitis)
* Known diagnosis of an autoimmune disease (e.g. hypo- or hyperthyroidism, celiac disease, rheumatoid arthritis)
* Known diagnosis of cystic fibrosis
* Known diagnosis of porphyria
* Current use of drugs which influence gastrointestinal motility, such as erythromycin, azithromycin, butyl scopolamine, domperidone, peppermint oil capsules, and Iberogast
* Known pregnancy or current lactation
* Condition leading to profound immunosuppression (HIV, infectious diseases leading to immunosuppression, bone marrow malignancies/use of systematic chemotherapy)
* Life expectancy < 12 months
* Use of concomitant medication, including proton pomp inhibitors (PPI), with the exception of pain medication (pain medication in the form of Paracetamol or NSAIDs is allowed)
* Use of systemic antibiotics in preceding 6 weeks
* Use of probiotic treatment in preceding 6 weeks
* Positive stool cultures for Clostridium difficile, Helicobacter pylori
* Positive Dual Faeces Test for Giardia lamblia, Dientamoeba fragilis, Entamoeba histolytica
* XTC, amphetamine or cocaine abuse
* History of surgery (hemicolectomy (defined as: surgery resulting in a resection of > 0.5 of the colon), presence of a pouch due to surgery, presence of stoma)
* Known intra-abdominal fistula
* Vasopressive medication, ICU stay
* Signs of ileus, diminished passage
* Allergy to macrogol or substituents, e.g. peanuts, shellfish
* Insufficient knowledge of the Dutch language

Donors

* Abnormal bowel motions, abdominal complaints or symptoms indicative of irritable bowel syndrome
* An extensive travel behaviour
* Unsafe sex practice (questionnaire)
* Use of any medication including PPI
* Antibiotic treatment in the past 12 weeks
* A positive history/clinical evidence for inflammatory bowel disease (Crohns disease or ulcerative colitis) or other gastrointestinal diseases, including chronic diarrhoea or chronic constipation
* A positive history/clinical evidence for autoimmune disease (type 1 diabetes, Hashimoto hypothyroidism, Graves hyperthyroidism, rheumatoid arthritis, celiac disease) and/or patients receiving immunosuppressive medications
* History of or present known malignant disease and/or patients who are receiving systemic anti-neoplastic agents
* Known psychiatric disease (depression, schizophrenia, autism, Asperger's syndrome)
* Known chronic neurological/neurodegenerative disease (e.g. Parkinson's disease, multiple sclerosis)
* Predisposing factors for potential transmittable diseases (e.g. regular sexual contact with prostitutes/promiscuity)
* Positive blood tests for the presence of: HIV, HTLV, lues, Strongyloides, amoebiasis
* Active hepatitis A, B-, C- or E-virus infection or known exposure within recent 12 months, acute infection with cytomegalovirus (CMV) or Epstein-Barr virus (EBV)
* Positive faecal tests for the presence of:

  * Bacteria (Clostridium difficile, Helicobacter pylori, Salmonella spp., Shigella spp., pathogenic Campylobacter spp., Yersinia enterocolitica, Aeromonas spp., Plesiomonas shigelloides, Antibiotic resistant bacteria: Extended spectrum beta-lactamase (ESBL)-producing Enterobactereacceae, VRE (vancomycin resistant enterococ)
  * Viruses (faecal PCR-test: Norovirus Type I and II, Astrovirus, Sapovirus, Adenovirus type 40/41, Rotavirus, Enterovirus, Adenovirus non-41/41)
  * Parasites (Giardia lamblia, Cryptosporidium spp., Entamoeba histolytica, Dientamoeba fragilis, Microsporidium spp., Blastocystis hominis, Isospora spp. Or more than 1 of the following non-pathogenic parasites: Entamoeba gingivalis, Entamoeba hartmanni, Entamoeba coli, Entamoeba polecki, Endolimax nana, Iodamoeba bütschlii, Entamoeba dispar, Entamoeba moshkovskii
* If a donor turns out positive for only 1 of the above mentioned non-pathogenic parasites, inclusion is acceptable

  o Parasitic worm eggs, larvae, protozoan cysts and oocysts
* Chronic pain syndromes (e.g. fibromyalgia)
* Major relevant allergies (e.g. food allergy, multiple allergies)
* Recent (gastrointestinal) infection (within last 6 months)
* Tattoo or body piercing placement within last 6 months
* Known risk of Creutzfeldt Jacobs disease
* History of current use of IV drugs
* History of treatment with growth factors
* Untreated infection with: Treponematoses, TBC, Herpes virus

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-11-23 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with > 50% reduction of their abdominal pain intensity and pain frequency at t=12 weeks after the first faecal transplantation | T=12 weeks
  This will be assessed with the pain component of the Irritable Bowel Syndrome Severity Scoring System (IBS-SSS) score. With 2 questions, the severity and frequency of the abdominal pain on the last 10 days is measured. The IBS-SSS is the only symptom severity scale that has been responsive to treatment effects. It has been recommended as the best instrument to obtain information on specific IBS related symptoms.

SECONDARY OUTCOMES:
Intra-individual changes in faecal gut microbiota composition | At baseline, 6 weeks, 12 weeks, 6 months and 12 months after faecal transplantation
  To examine the changes in faecal microbiota composition in IBS patients following FMT. To assess faecal gut microbiota composition, morning stool samples will be collected. Samples will be taken by the patient him/herself (wearing gloves) and will be put in a small container. Afterwards it will directly be transported to the AMC, where all samples will be stored at -80°C. Faecal analysis will be done by HITChip flora mapping, an established sensitive RT-qPCR method which is developed for exact and sensitive enumeration of bacterial population.
Adverse events | At t=3, t=6, t=12 and t=16 weeks, and t=6 and 12 months
  Participants will be screened for adverse events from the time of informed consent through the end of the trial. In case of an identified adverse event, this will be recorded and described in the CRF.
The proportion of patients with > 50% reduction of their abdominal pain intensity and pain frequency | At t=6 and t=12 months
  This will be assessed with the pain component of the Irritable Bowel Syndrome Severity Scoring System (IBS-SSS) score.
Total IBS-SSS score | At baseline, t=3, t=6, t=12 and t=16 weeks, and t=6 and 12 months
  In addition to the pain component of the IBS-SSS score, the total IBS-SSS score will be evaluated with the same interval.
Health related quality of life | baseline, t=6 and t=12 weeks, and t=6 and 12 months
  The IBS-QOL questionnaire will be used as the disease specific questionnaire. This questionnaire is a 34-item assessment of the degree to which the IBS interferes with patient quality of life and consists of eight domains: dysphoria, interference with activities, body image, health worry, food avoidance, social reactions, sexual health, and effect on relationships. For generic quality of life, the Medical Outcomes Study 36-item Short Form Health Survey (SF-36) will be used.The SF-36 questionnaire consists of 36 questions regarding eight dimensions of health perception: limitations in physical functioning, role limitation due to physical health problems, bodily pain, general health perception, vitality, social functioning, role limitations due to emotional limitations, and mental health. The reliability has been proven extensively for diverse patient groups and it is validated for the Dutch population.The SF-36 is described as adequate for persons 14 years of age and older.
Depression and anxiety | baseline, t=6 and t=12 weeks, and t=6 and 12 months.
  Depression and anxiety scores will be measured using the SCL-90. The SCL-90 is a widely used measure of psychological state, suitable for adolescents > 11 years and adults. It has question items that ask on a 5-point scale, how much a certain problem has bothered the subject over the past 7 days. This allows nine scales to be derived, namely somatisation, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism
Absence of school or work, health care resources and costs | baseline, t=6 and t=12 weeks, and t=6 and 12 months.
  A self-designed questionnaire will be used to monitor school absence (adolescents) and absence from work during the first year after treatment.
Adequate relief | t=6 and t=12 weeks, and t=6 and 12 months
  Adequate relief will be measured using a single question ("Did you have adequate relief of IBS/FAP symptoms (abdominal discomfort/pain, bowel habits, and other symptoms like nausea and bloating) over the past week?") scored on a dichotomous scale (Yes/No). This instrument is a well-validated simple outcome assessment for IBS treatment.
Number of participants with treatment-related adverse events as assessed by CRP, liver profile and renal profile | t=0, t=6 and t=12 weeks
  CRP, liver profile and renal profile will be assessed.Therefore, 4 tubes of blood per assessment will be taken, with a total maximum amount of 20mL. Three of these tubes will be frozen and stored. In case certain biomarkers for inflammation or metabolites related to the gut-brain axis will be demonstrated in the next 5 years, the stored serum can be used for analysis of this newly discovered biomarkers or metabolites in irritable bowel syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Benninga, Prof.dr, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeevenhooven J, de Bruijn CMA, Vlieger A, Nieuwdorp M, Benninga MA. Protocol for a pilot randomised, double-blind, placebo-controlled trial for assessing the feasibility and efficacy of faecal microbiota transplantation in adolescents with refractory irritable bowel syndrome: FAIS Trial. BMJ Paediatr Open. 2020 Aug 20;4(1):e000689. doi: 10.1136/bmjpo-2020-000689. eCollection 2020. PMID 32864480